CLINICAL TRIAL: NCT05987709
Title: Study of Colorectal Cancer Screening Options
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: KPNW Guardant [1866832-1]
Record Dates: First submitted 2023-07-07; First posted 2023-08-14 (Actual); Results first posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Colon Cancer
Keywords: Colon Cancer Screening
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guardant Shield Blood Test (Other): Patients will have the Guardant Shield blood test for colorectal cancer screening.
  Interventions: Diagnostic Test: GuardantSHIELD Blood Test
- Standard of Care (No Intervention): Patients will have standard of care, which is a reminder to do their FIT test for colorectal cancer screening

INTERVENTIONS:
Diagnostic Test: GuardantSHIELD Blood Test — The GuardantSHIELD CRC screening test is a commercially available test which works by finding signs of colorectal tumor in the blood of patients at average risk for CRC
  Arms: Guardant Shield Blood Test

SUMMARY:
The investigators propose to evaluate Guardant Health's commercially available colorectal cancer screening assay(Guardant SHIELD) in individuals who are not up to date with CRC screening.

DETAILED DESCRIPTION:
The investigators propose to evaluate Guardant Health's commercially available colorectal cancer screening assay(Guardant SHIELD) in individuals who are not up to date with CRC screening.

Primary Objective (or Aim) Assess colorectal cancer screening completion among patients who are non-adherent after receiving stool test outreach, who have an upcoming clinical appointment, and who are offered a commercially available colorectal cancer blood test versus usual care (i.e. reminder to complete stool testing during their clinical appointment).

Secondary Objectives (or Aim) Assess patients' and providers' perceived confidence in the test (based on available test performance characteristics) and willingness to obtain/offer the test on an on-going basis, based on qualitative interviews; assess preliminary rates of follow-up colonoscopy completion (after an initial abnormal test result) among participants allocated to the blood test vs. usual care condition.

ELIGIBILITY:
Inclusion Criteria:

* Age 45-75
* Received a FIT test in the last 3-9 months yet did not return their FIT
* Upcoming appointment or willing to reschedule an appointment at KPNW within 2 - 6 weeks
* Able and willing to provide informed consent if in the intervention arm

Exclusion Criteria:

* On KPNW's do not contact list
* Having a legal authorized representative
* Non-English speakers

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2004 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Coronado, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Northwest, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Coronado GD, Jenkins CL, Shuster E, Johnson C, Amy D, Cook J, Sahnow S, Zepp JM, Mummadi R. Blood-based colorectal cancer screening in an integrated health system: a randomised trial of patient adherence. Gut. 2024 Mar 7;73(4):622-628. doi: 10.1136/gutjnl-2023-330980. PMID 38176899

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Guardant Shield Blood Test | Standard of Care
Started | 1001 | 1003
Completed | 1001 | 1003
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Guardant Shield Blood Test | Standard of Care | Total
Number analyzed (Participants) | 1001 | 1003 | 2004
Age, Customized [Count of Participants; unit: Participants]
  45-49 | 29 | 28 | 57
  50-64 | 718 | 722 | 1440
  65-75 | 254 | 253 | 507
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 642 | 598 | 1240
  Male | 359 | 405 | 764
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 45 | 31 | 76
  Black | 60 | 55 | 115
  Hispanic(any race) | 31 | 35 | 66
  Other/Multiple/Unknown | 73 | 73 | 146
  White | 792 | 809 | 1601
Prior CRC Screening [Count of Participants; unit: Participants]
  Prior CRC Screening | 521 | 520 | 1041
  No Prior CRC Screening | 480 | 483 | 963

OUTCOME MEASURES:

1. Primary Outcome: Assess Colorectal Cancer Screening Completion
Description: Assess the percentage who received any CRC screening test (blood draw, FIT or FIT-DNA, or flexible sigmoidoscopy or colonoscopy) within 3 months of eligibility determination among eligible individuals in the blood test and usual care groups.
Time Frame: Within 3 months of patient identification
Measure: Count of Participants; unit: Participants
Arm/Group | Guardant Shield Blood Test | Standard of Care
Number analyzed (Participants) | 1001 | 1003
Participants | 305 | 130

2. Secondary Outcome: Assess the Percentage of Participants Who Completed Follow-up Testing.
Description: Assess the percentage of participants who completed follow-up colonoscopy within 6 months of their result among individuals with an abnormal non-invasive test result; comparing the blood test and usual care groups.
Time Frame: Within 6 months of abnormal FIT test
Measure: Count of Participants; unit: Participants
Arm/Group | Guardant Shield Blood Test | Standard of Care
Number analyzed (Participants) | 22 | 10
Participants | 11 | 7

ADVERSE EVENTS:
Time Frame: 9 Months
Arm/Group | Guardant Shield Blood Test | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/1001 | 0/1003
Serious Adverse Events (participants affected / at risk) | 0/1001 | 0/1003
Other Adverse Events (participants affected / at risk) | 1/1001 | 0/1003
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Guardant Shield Blood Test (N=1001) | Standard of Care (N=1003)
Pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Patient had continued pain at site of the blood draw, the "puncture wound" would not stop hurting. Patient got care at an urgent care, no treatment necessary

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2022-10-07): https://cdn.clinicaltrials.gov/large-docs/09/NCT05987709/Prot_ICF_000.pdf